CLINICAL TRIAL: NCT02394847
Title: Does Repetitive Electroconvulsive Therapies Affect Propofol Induction Dose?
Brief Title: Does Repetitive Electroconvulsive Therapies Affect Propofol Induction Dose ?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, CIGDEM YILDIRIM GUCLU, specialist anesthesiologist, Ankara University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 14835
Record Dates: First submitted 2015-03-08; First posted 2015-03-20 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Physiatrics; Electroconvulsive Therapy
Keywords: propofol; electroconvulsive therapy; anesthesia
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- propofol (Other): dose of propofol according to the number of therapies
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol

SUMMARY:
Electroconvulsive therapy has been used for many years for different types of physiatric diseases. General anesthesia is used during the procedure. Different anesthesiologists use different regimens. The duration of seizure is important in this procedure. The investigators evaluated the relationship between the dose of propofol and the number of electroconvulsive therapy and duration of the seizure.

ELIGIBILITY:
Inclusion Criteria:

* Patients required electroconvulsive therapy for the physiatric disease

Exclusion Criteria:

* Patients refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
dose of propofol | 10 seconds

SECONDARY OUTCOMES:
duration of seizure | 10 seconds